CLINICAL TRIAL: NCT06252571
Title: a Chronobiological Treatment Combining Evening Melatonin and Morning Light Therapy in Idiopathic Hypersomnia: a Prospective, Double Bind, Randomized, Placebo-controlled -Trial
Acronym: HyperChrono
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 8443
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Idiopathic Hypersomnia
Keywords: hypersomnia; light; melatonin; sleep; chronobiotherapy
MeSH Terms: conditions — Idiopathic Hypersomnia; Disorders of Excessive Somnolence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active therapy (Experimental): Active therapy combining evening melatonin + morning active light over 6 weeks
  Interventions: Combination Product: - Melatonin - Active light ttherapy
- Placebo therapy (Placebo Comparator): placebo therapy combining evening melatonin placebo + morning placebo light over 6 weeks.
  Interventions: Combination Product: - Placebo drug - Placebo light therapy

INTERVENTIONS:
Combination Product: - Melatonin - Active light ttherapy — 1 tablet per day, in the evening + morning light therapy over 6 weeks
  Arms: Active therapy
Combination Product: - Placebo drug - Placebo light therapy — 1 tablet per day in the evening + morning placebo light therapy
  Arms: Placebo therapy

SUMMARY:
Idiopathic hypersomnia (IH) is a chronic disabling disorder characterized by excessive daytime sleepiness (EDS), prolonged nighttime sleep and sleep inertia. IH is a rare disorder, estimated around 0.05%, yet its true prevalence remains unknown. Disease onset occurs most often during young adulthood and is accompanied by severe social, professional and economic impairments, resulting in risk of accident and a loss in patient's quality of life. There are no ANSM (or FDA-) approved treatments for IH symptoms.

IH shares common features with delayed sleep-wake phase disorder (DSWPD) which is a chronic circadian rhythm disorder which occurs as in IH during young adulthood. The combination of evening melatonin and morning bright light therapy is the most effective validated chronotherapy in DSWPD.Moreover, bright light therapy has direct effects and is known to increase daytime alertness and to improve mood.

Melatonin is empirically used in routine clinical practice in patients with IH and French and European recommendations mention melatonin as a possible treatment of sleep inertia in IH.

. Our goal is to bring a proof of concept of a safe therapeutic practice for IH combining exogenous melatonin and bright light therapy in

ELIGIBILITY:
Inclusion criteria:

* Male or female patient
* Age ≥ 18 and ≤ 40 years at signature of informed consent form
* Diagnosed with Idiopathic hypersomnia in a reference/competence center of hypersomnia rare disease network according to ICSD-3 criteria (International classification of sleep disorders) with symptoms lasting since >3 months and a total sleep time ≥11hours objectified with a 24h continuous polysomnography realized during the last 12 months
* Patient with stable medication in the month preceding inclusion and throughout the 10 weeks of participation to the study (except for drugs excluding participation. See list below).
* Patient able to be compliant with therapy during the required time and at the set schedule.
* For female patient: effective efficient contraception during the month preceding the inclusion and all along the study
* Patient who have given written informed consent and are able to understand the objectives and risks associated to the research.
* Patient affiliated to a social security insurance

Exclusion criteria:

1. Criteria related to the underlying disorder (other forms of hypersomnia or sleep disorder)

   * Other primary or secondary hypersomnia (narcolepsy, Kleine-Levin syndrome, post-traumatic hypersomnia, hypersomnia due to medication or substance abuse…)
   * Other intrinsic sleep disorder according to ICSD-3 criteria (sleep apnea syndrome, restless legs syndrome, insomnia)
2. Criteria related to pathologies associated with particular risks or consumption of substances that may affect sleep or alertness:

   * Significant psychiatric comorbidities (current severe depressive episode based on the DSM-V criteria, risk of suicide, schizophrenia, bipolar disorder).
   * Known systemic or severe acute disease (auto-immune diseases…)
   * Substance / alcohol /cigarette dependence
   * Consumption of excessive amounts of caffeine, defined as greater than 600 mg of caffeine of coffee, tea, cola, energy drinks, or other caffeinated beverages per day (1 cup of coffee is approximately 120 mg)
3. Criteria related to circadian rhythms disturbances

   * Recent transmeridian travel (> 2 time zones) within the month before the start of the study
   * History of shift/night work reported within the 6 months preceding the study
   * Irregular sleep habits (more than 2 hours of delay or advance in bedtime ≥ 3 nights over a week)
   * Circadian sleep-wake rhythm disorders according to ICSD-3 criteria (advanced or delayed sleep phase syndrome, …)
4. criteria related to medications (within 1 month prior to study)

   * Sleep promoting drugs (benzodiazepines, z-drugs, sodium oxybate, antihistaminics…)
   * Wake promoting-drugs (modafinil, pitolisant, methylphenidate, solriamfétol chlorhydrate)
   * Psychotropics and drugs inducing level 3 sleepiness according to the ANSM (French National Agency for Medicines and Health Products Safety) gradation.
   * beta-blockers
   * regular anti-inflammatory drug intake
   * Exogenous melatonin and/or serotonin and or tryptohane (as a drug or a dietary supplement)
5. Criteria related to relative contra-indications to light therapy

   * Medical history of ophthalmologic diseases causing visual impairment: retinopathy, age-related macular degeneration, macular hole, epiretinal membrane; cataract; optic neuropathy.
   * On-going medication with a photosensibilizing drug
   * Photosensitive epilepsia or migraine
6. Criteria relative to exogenous melatonin administration

   * Prior intolerance to cellulose or exogenous melatonin
   * Drugs metabolized by CYP1A2 intake within 1 month prior to study: antivitamin K, fluvoxamine, cimetidine, carbamazepine, rifampicin…
7. Criteria relative to relative contraindications of e-celsius capsules

   * Patient weighting less than 40 kg
   * Medical history of motility disorders of the gastrointestinal tract and intestinal disorders that can lead to obstruction of the digestive tract, including diverticula, Crohn disease, surgical procedures in the gastrointestinal tract
   * Known swallowing disorders
   * In presence of a pacemaker or electro-medical implant.
   * Patient who has to undergo strong electromagnetic field during the period of use of the system (MRI)
8. Criteria relative to regulation:

   * Pregnancy, breastfeeding.
   * Participation in another interventional clinical trial with an exclusion period
   * Patient with difficulty to read or understand French, or inability to understand the delivered information
   * Patient in emergency situation
   * Patient in life-threatening situation
   * Patient under justice safeguard
   * Patient under guardianship or limited guardianship
   * Patient unwilling to refrain from driving and/or operating dangerous or hazardous machinery during times of heightened sleepiness or fatigue due to the medication

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-09-07 (Actual); Primary Completion 2027-09-07 (Estimated); Study Completion 2027-09-07 (Estimated)

PRIMARY OUTCOMES:
Idiopathic Hypersomnia Severity Severity Scale (IHSS) | At Day 14 and day 45
  The Idiopathic Hypersomnia Severity Severity Scale is a self-administered questionnaire that was designed specifically to quantify HI symptoms the minimum value is 0 and the maximum values 50 means a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No